CLINICAL TRIAL: NCT04586933
Title: Nutritional Intervention in Rheumatic Diseases: Effect of Marine Omega-3 Fatty Acids and Individual Dietary Guidance
Brief Title: Nutrition in Rheumatic Diseases
Acronym: EROM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haukeland University Hospital (Other)
Collaborators: GC Rieber Oils AS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 79907
Record Dates: First submitted 2020-09-22; First posted 2020-10-14 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Spondyloarthritis; Rheumatoid Arthritis; Polyarthritis
Keywords: Fatty acids; Diet; Nutritional Status
MeSH Terms: conditions — Spondylarthritis; Arthritis, Rheumatoid; Arthritis | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Intervention Model Description: The study will be twofold and consist of Intervention 1 and Intervention 2.
  Intervention 1: Dietary guidance (12 weeks). All participants will receive individual dietary guidance, as well as an intensive dietary course with 4 sessions. Participants will receive contact information to the clinical dietitian, and the opportunity to ask questions throughout the intervention period. Patients will be asked to not use other omega-3 supplement during the intervention period 1.
  Intervention 2: Omega-3 vs. placebo (24 weeks). After intervention 1, patients will be randomized to take either 3 grams of omega-3 or placebo daily, divided into 4 capsules. Patients will be asked not to use other omega-3 supplements in the period from 2 months until after intervention period 2.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega-3 (Active Comparator): 0,9 gram omega-3/capsule x 4 = 3,6 gram omega-3 daily
  It will be investigated whether diet optimization followed with supplementation of omega-3s can reduce disease activity in patients with inflammatory arthritis. A new omega-3 high concentrate from GC Rieber Oils will be used
  Interventions: Dietary Supplement: Omega-3; Behavioral: Dietary guidance
- Placebo capsules (Placebo Comparator): Soya oil
  Interventions: Dietary Supplement: Placebo (soya); Behavioral: Dietary guidance

INTERVENTIONS:
Dietary Supplement: Omega-3 — It will be investigated whether diet optimization and supplementation of omega-3s can reduce disease activity in patients with inflammatory arthritis. A new omega-3 high concentrate from GC Rieber Oils will be used.
  Arms: Omega-3
Dietary Supplement: Placebo (soya) — Placebo (soya)
  Arms: Placebo capsules
Behavioral: Dietary guidance — Dietary guidance

SUMMARY:
Background: Patients with inflammatory rheumatic diseases (IRD) are prone to malnutrition for several reasons. The diseases and treatment can cause reduced intake and absorption of nutrients and the inflammatory processes may cause an increased demand for nutrients, especially proteins. Studies report that nutritional status can affect disease activity. Dietary supplement of 3-4 gram omega-3 has shown beneficial effect upon disease activity in patients with IRD.

Aim: To investigate whether improved dietary intake with and without supplements of omega-3 will affect disease activity in patients with rheumatoid arthritis (RA) and spondyloarthritis (SpA).

Hypothesis 1: A systematic change of diet in line with the Norwegian dietary guidelines, which will result in increased intake of, among other nutrients, omega-3 fatty acids and complete protein, as well as reduced intake of saturated fat and sugar, will improve nutritional status and reduce disease activity.

Hypothesis 2: A systematic change of diet (as above), included a high dose of omega-3 will further improve nutritional status and reduce disease activity compared with placebo.

Design: A DB-RCT-study will be conducted. All patients will receive individualized dietary guidance by a clinical dietician for 12 weeks, before randomization to supplements of omega-3 or placebo, for 24 weeks. The supplement will be blinded for the participants, researchers and physicians.

Clinical implications: The study will investigate the effect of improved diet and nutrition on treatment offered to patients with IRD to provide more evidence-based knowledge, and thus specific dietary guidelines for patients with IRD. In addition, the study might increase the understanding of the role of omega-3 in the pathogenesis of inflammation.

DETAILED DESCRIPTION:
The study is approved by the Regional Committee for Medical and Health Research Ethics. Participation is voluntary, and informed consent will be requested. Outpatients will be recruited by doctors at the Rheumatology Department at Haukeland University Hospital (HUH). Patients recruited will be included consecutively. The recruitment period will last up to 12 months. Anthropometrical measurements, analysis of body composition, blood tests, clinical parameters, and dietary data will be collected at baseline, and after 12, 24, 36 and 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed with one of the following diagnoses: rheumatoid arthritis, according to the ACR / EULAR 2010 criteria, psoriatic arthritis, according to the CASPAR criteria, axial spondylarthritis, including ankylosing spondylarthritis and non-radiographic spondylarthritis, according to the ASAS criteria
* Duration of illness ≥0.5 years
* Between 18 and 75 years
* Understand Norwegian
* The patient has given informed consent to participate
* No change in medication the last 12 weeks before inclusion

Exclusion Criteria:

Diagnoses / conditions that make it difficult to follow a dietary intervention and / or supplementation of omega-3s, including:

* Conditions or use of medications where omega-3 is contraindicated
* Pregnancy / lactation
* Allergy to soy or fish
* Severe liver disease
* Severe mental or physical illnesses, such as insulin-requiring diabetes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2025-06-10 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
DAS28 (Disease Activity Score 28-joint count) | Change between week 0, 12, 24, 36 and 52
  Disease activity score, higher values indicate a higher disease activity and below 2.6 meaning remission.
ASDAS-CRP (Ankylosing Spondylitis Disease Activity Score) | Change between week 0, 12, 24, 36 and 52
  Disease activity score, higher values indicate a higher disease activity
DAPSA (Disease Activity Index for Psoriatic Arthritis) | Change between week 0, 12, 24, 36 and 52
  Disease activity score, higher values indicate a higher disease activity and below 4 meaning remission

SECONDARY OUTCOMES:
RAID (Rheumatoid Arthritis Impact of Disease) | Change between week 0, 12, 24, 36 and 52
  Disease activity scores and scores evaluating quality of life, range 0-10, and higher scores indicate a higher grade of disability
RAND12 (short form health survey) | Change between week 0, 12, 24, 36 and 52
  Disease activity scores and scores evaluating quality of life
MHAQ (Modified Health Assessment Questionnaire) | Change between week 0, 12, 24, 36 and 52
  Disease activity scores and scores evaluating quality of life, range from 0 to 3 while higher values indicate a higher grade of disability
BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) | Change between week 0, 12, 24, 36 and 52
  Disease activity scores and scores evaluating quality of life, range 0-10, and higher values indicate higher disease activity
BASFI (Bath Ankylosing Spondylitis Functional Index) | Change between week 0, 12, 24, 36 and 52
  Disease activity scores and scores evaluating quality of life, range 0-10, and higher values indicate a higher grade of disability
CDAI (Clinical Disease Activity Index) | Change between week 0, 12, 24, 36 and 52
  Disease activity scores and scores evaluating quality of life, range 0-76, and scores below 2.8 indicate remission
Consumption of medicine after 12 months | Change between baseline and week 52
  The proportion who must start or change biological treatment, use of NSAIDs and steroids
BMI (Body Mass Index) | Change between week 0, 12, 24, 36 and 52
  Nutritional status: Weight (kg) and height (m) will be combined to report BMI (kg/m^2) Change in BMI, waist circumference, fat mass (kg), fat-free mass (kg), fat-free mass index (kg/m2), fat-mass index (kg/m2), handgrip strength
Waist circumference | Change between week 0, 12, 24, 36 and 52
  Nutritional status: Waist circumference (cm)
Handgrip strength | Change between week 0, 12, 24, 36 and 52
  Nutritional status: Handgrip strength, measured by a dynamometer (kg)
Body composition | Change between week 0, 12, 24, 36 and 52
  Estimation of fat mass (kg), fat-free mass (kg), measured by BIA and DXA. Fat-free mass index (kg/m2), and fat-mass index (kg/m2) will be calculated.
Dietary intake of macro- and micronutrients, based on a dietary registration of 7 days | Week -1,10, 50
  Energy (E%, kcal) proteins (g and E%) ratio of fatty acids fibers (g) Vitamins and minerals
Dietary intake of macro- and micronutrients, based on a 24h recall. | Week 0, 12, 24, 36, 52
  Energy (E%, kcal) proteins (g and E%) ratio of fatty acids fibers (g) Vitamins and minerals
Blood lipid profile | Change from week 0, 12, 24, 36 and 52
  HDL (mmol/L) LDL (mmol/L) total cholesterol (mmol/L) triglycerides (mmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Kristine H Halse, MD, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in articles will be shared, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available from 9 months and ending 36 months following article publication.
Access Criteria: IPD will be shared with investigators who provide a methodologically sound proposal, and whose use of data has been approved by a Human Subjects Protection Review Board.
  Proposal can be directed to marienjerve@gmail.com